CLINICAL TRIAL: NCT04858373
Title: Characterizing the Technological Properties of Emmer Seeds, Flour, and Bread; and Determining the Effect of Emmer Breads on Glycemic Responses in Healthy Humans
Brief Title: Characterizing Emmer Seeds and Flours, and Determining the Glycemic Effects of Emmer Breads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HRBD 39 12/07/2019
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; emmer bread; glycemic index; glycemic load; blood pressure
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glucose as reference food (Experimental): Fourteen healthy, normal weight subjects (male: 6, female: 8) after 12hr fast, consumed 50g available carbohydrates from D-glucose, three times, in different visits as reference food along with 300ml water; and 50g available carbohydrates from emmer bread from Greek emmer seeds, emmer bread from Italian emmer seeds, and whole wheat commercial soft bread, tested once, in different visits. there was a washout period of 2 days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Emmer bread from Greek emmer; Other: Emmer bread from Italian emmer; Other: Whole wheat commercial bread
- Emmer bread from Greek emmer (Experimental): Fourteen healthy, normal weight subjects (male: 6, female: 8) after 12hr fast, consumed 50g available carbohydrates from D-glucose, three times, in different visits as reference food along with 300ml water; and 50g available carbohydrates from emmer bread from Greek emmer seeds, emmer bread from Italian emmer seeds, and whole wheat commercial soft bread, tested once, in different visits. there was a washout period of 2 days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Emmer bread from Greek emmer; Other: Emmer bread from Italian emmer; Other: Whole wheat commercial bread
- Emmer bread from Italian emmer (Experimental): Fourteen healthy, normal weight subjects (male: 6, female: 8) after 12hr fast, consumed 50g available carbohydrates from D-glucose, three times, in different visits as reference food along with 300ml water; and 50g available carbohydrates from emmer bread from Greek emmer seeds, emmer bread from Italian emmer seeds, and whole wheat commercial soft bread, tested once, in different visits. there was a washout period of 2 days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Emmer bread from Greek emmer; Other: Emmer bread from Italian emmer; Other: Whole wheat commercial bread
- Whole wheat commercial bread (Experimental): Fourteen healthy, normal weight subjects (male: 6, female: 8) after 12hr fast, consumed 50g available carbohydrates from D-glucose, three times, in different visits as reference food along with 300ml water; and 50g available carbohydrates from emmer bread from Greek emmer seeds, emmer bread from Italian emmer seeds, and whole wheat commercial soft bread, tested once, in different visits. there was a washout period of 2 days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Emmer bread from Greek emmer; Other: Emmer bread from Italian emmer; Other: Whole wheat commercial bread

INTERVENTIONS:
Other: Glucose as reference food — Fourteen healthy, normal weight subjects (male: 6, female: 8) after 10-14 hr fast, consumed 50g glucose diluted in 300ml water, tested three times, in different visits, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Emmer bread from Greek emmer — Fourteen healthy, normal weight subjects (male: 6, female: 8) after 10-14 hr fast, consumed 50g available carbohydrates from Greek emmer bread, tested once, in different visits, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Emmer bread from Italian emmer — Fourteen healthy, normal weight subjects (male: 6, female: 8) after 10-14 hr fast, consumed 50g available carbohydrates from Italian emmer bread, tested once, in different visits, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Whole wheat commercial bread — Fourteen healthy, normal weight subjects (male: 6, female: 8) after 10-14 hr fast, consumed 50g available carbohydrates from whole wheat commercial bread, tested once, in different visits, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.

SUMMARY:
This study characterized emmer seeds, flours, and breads, and investigated the effects of emmer breads on the glycemic response

DETAILED DESCRIPTION:
This study aimed to 1. describe the technological characteristics of emmer seeds, flours, and breads, 2. determine the glycemic index and glycemic load of two emmer breads, and 3. to investigate the effects of these breads on postprandial glycemic response in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* non-diabetic men and women
* body mass index (BMI) between 18 and 27 kg/m2

Exclusion Criteria:

* severe chronic disease (e.g. coronary heart disease, diabetes mellitus,kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol
* drug dependency

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet,one scale per page) at baseline, 15, 30, 45, 60, 90 and 120 min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g hunger, satiety, desire to eat etc.
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2hr after consumption of the breads

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece